CLINICAL TRIAL: NCT06655454
Title: The Effects of Supplemental Postoperative 0.5% Bupivacaine With 1:200,000 Epinephrine Following Non-Surgical Endodontic Treatment on Patients' Quality of Life, Pain, and Analgesic Consumption
Brief Title: Supplemental Postoperative Bupivacaine Following Non-Surgical Endodontic Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: i24-01018
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-11

CONDITIONS: Pain Assessment; Quality of Life (QOL); Analgesic Use
Keywords: bupivacaine; nonsurgical endodontic treatment; root canal therapy; irreversible pulpitis; pain management; anesthetic use
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Three types of additional treatment after standard nonsurgical endodontic procedures may be given. These include an additional injection of bupivacaine, an additional mock or placebo injection, and no additional injection.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Supplemental Postoperative Bupivacaine (Experimental): An additional injection, 1 carpule (1.8 mL) of 0.5% bupivacaine with 1:200,000 epinephrine, will be given to patients in this treatment arm, after their standard endodontic procedure is complete.
  Interventions: Drug: Supplemental Postoperative Bupivacaine
- Mock/Placebo Injection (Placebo Comparator): If assigned to this arm, the patient will be shown the removal of a needle cap for an anesthetic syringe. The tip will be bent and placed in the patient's mouth, but no tissue penetration will occur. No solution of anesthetic will be delivered.
  Interventions: Drug: Placebo Injection
- No Additional Injection (No Intervention): After standard endodontic procedure, no additional injection will be given.

INTERVENTIONS:
Drug: Supplemental Postoperative Bupivacaine — This is the intervention of interest. A supplemental injection of bupivacaine will be given postoperatively to patients who are assigned this intervention.
  Arms: Supplemental Postoperative Bupivacaine
Drug: Placebo Injection — This intervention will appear to give patients an additional injection, but no additional drug will be given.
  Arms: Mock/Placebo Injection

SUMMARY:
The study will investigate the impact of an additional injection of long-acting anesthetic on pain level, quality of life, and use of pain medication after a nonsurgical endodontic treatment. The long-acting anesthetic will be compared to a mock injection group and a group with no additional anesthetic to determine any differences in effects.

DETAILED DESCRIPTION:
The study will investigate the impact of postoperative supplemental long-acting bupivacaine on patient's pain, quality of life, and analgesic use following treatment for symptomatic irreversible pulpitis on patients with pre-operative pain levels of 5 or above (on a 0-10 analog scale). Bupivacaine will be compared to a placebo/mock injection and no injection to determine the difference in effect.

ELIGIBILITY:
Inclusion Criteria:

1. Medical ASA Class I or II
2. Patients above 18 years old
3. Patients with a blood pressure below 160/100
4. Patients who are treatment planned and have agreed to have emergency endodontic therapy or non-surgical root canal therapy with a pulpal diagnosis of symptomatic irreversible pulpitis according to the AAE Glossary of Endodontic Terms.
5. Patients must be able to comprehend and complete all study protocols, written consent, and questionnaires in English.

Exclusion Criteria:

1. Medical ASA III or above
2. Patients who reported the use of tobacco or nicotine-containing products such as vapes, e-cigarettes, gums, or pouches and will not in the 48 hours following treatment
3. Patients who reported the use of any marijuana products or illicit drugs in the 48 hours prior to treatment and will not in the next 48 hours.
4. Patients who have taken opioids to control pain.
5. Pregnant patients
6. Patients with a blood pressure of 160/100 or greater
7. Patients with a known hypersensitivity or allergy to any local anesthetic agent of the amide group, or any other components of the two anesthetic solutions such as epinephrine, sodium metabisulfite used in the study.
8. Patients who have more than one tooth with odontogenic pain at the time of the screening.
9. Patients who are unable to consent and do not understand or are unable to read the questionnaires.
10. Patients who have had 4 1.7 ml carpules or more of anesthetic (Lidocaine and/ or Septocaine, 1:100,000) during standard care of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life | Day of operation and daily for four days immediately following endodontic treatment
  Quality of life will be measured with a modified version of the OHIP-14 questionnaire.
  For each question, the answers correspond with a scale that runs from 0-4. A higher score corresponds with a lower quality of life, with 0 being great quality of life and 4 being very poor quality of life.

SECONDARY OUTCOMES:
Postoperative pain level | Day of operation and daily for four days immediately following endodontic treatment
  Pain level as measured by the visual-analog scale (VAS) will be collected for four days following endodontic treatment.
  The scale is from 0-10, with 0 being no pain and 10 being the worst pain possible.
Analgesic use | Day of operation and daily for four days immediately following endodontic treatment
  Use of self-administered analgesics including opioids will be measured postoperatively.
  The measure is binary- either usage of self-administered analgesics or no usage of self-administered analgesics.

CONTACTS AND LOCATIONS:
Locations (1):
- New York University College of Dentistry, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No